CLINICAL TRIAL: NCT05808933
Title: Magnetic Resonance Fingerprinting for Preoperative Evaluation of Lymphovascular Space Invasion in Early Stage Cervical Cancer
Acronym: MARF-ESC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4988
Record Dates: First submitted 2023-03-06; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational prospective study is to investigate the role of Magnetic Resonance Fingerprinting in preoperative assessment of early cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven cervical cancer FIGO stage IA-IIA undergoing surgery;
* Women aged >18 years old;
* Signed Informed Consent.

Exclusion Criteria:

* Concurrent malignancies at other sites;
* Previous history of neoplasm;
* Refusal to sign written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of cervical cancer (FIGO IA-IIA) that will undergo to surgery at Fondazione Policlinico Universitario "A. Gemelli" IRCCS can be included in this study, according to inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Association between T1-, T2- and ADC-maps and LVSI status | 3 months

SECONDARY OUTCOMES:
Correlation between T1-, T2- and ADC-maps and DFS and OS | 3 years
Correlation between Radiomics-based analysis and LVSI status and DFS and OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy